CLINICAL TRIAL: NCT05629962
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Bemnifosbuvir in High-Risk Outpatients With COVID-19
Brief Title: SUNRISE-3: Efficacy and Safety of Bemnifosbuvir in High-Risk Outpatients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-03A-017
Record Dates: First submitted 2022-11-26; First posted 2022-11-29 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV 2 Infection); COVID-19
MeSH Terms: conditions — COVID-19 | interventions — AT-511

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bemnifosbuvir (BEM) (Experimental)
  Interventions: Drug: Bemnifosbuvir (BEM)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bemnifosbuvir (BEM) — BEM tablets administered orally every 12 hours (twice a day) for a total of 5 days
  Other Names: AT-527
  Arms: Bemnifosbuvir (BEM)
Drug: Placebo — Placebo tablets administered orally every 12 hours (twice a day) for a total of 5 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether bemnifosbuvir (BEM) is effective and safe in adults with COVID-19 who do not need to be in the hospital but who are at high risk for progression to severe disease. Eligible subjects will be randomly assigned (by chance) to receive BEM or matching placebo orally for 5 days. Co-administration of locally available standard of care (SOC) is allowed. The total duration of the study is 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 test conducted ≤ 5 days prior to randomization
* Mild or moderate COVID-19 with symptom onset ≤ 5 days before randomization and at least one COVID-19 related symptom present at time of screening
* Subject must be high risk, defined below:

  1. Age ≥70 years OR
  2. Age ≥55 years with one of the following: i) obesity (body mass index [BMI] ≥30 kg/m2) ii) diabetes mellitus iii) cardiovascular disease or hypertension iv) chronic lung disease requiring routine therapy OR
  3. Age 50 to 54 years with two of the following: i) obesity (BMI ≥30 kg/m2) ii) diabetes mellitus iii) cardiovascular disease or hypertension iv) chronic lung disease requiring routine therapy OR
  4. Age ≥18 years with one of the following: i) Down syndrome, sickle cell disease, dementia, Parkinson's disease, or care home residents ii) One of the following immunocompromising conditions or immunosuppressive treatments: receiving chemotherapy for cancer, hematologic malignancy, being within 2 years of a hematopoietic stem cell transplant, receipt of a solid organ transplant and on immunosuppressive therapy, human immunodeficiency virus (HIV) infection untreated or with CD4+ T lymphocyte count <350 cells per cubic millimeter, moderate/severe primary immunodeficiency, taking immunosuppressive medications
* Use of adequate contraception for females of childbearing potential

Exclusion Criteria:

* Severe or critical COVID-19 illness
* Admitted to a hospital within 90 days prior to randomization due to COVID-19
* Use of other investigational drugs within 30 days prior to planned dosing, or plans to enroll in another clinical trial of an investigational agent while participating in the present study
* Initiation or planned initiation of remdesivir for treatment of the current SARS-CoV-2 infection
* Requirement of prohibited medications, including hydroxychloroquine or amiodarone within 3 months prior to screening. Note: Subjects who had already initiated any COVID-19 drug with antiviral effects intended to treat symptomatic SARS-CoV-2 infection (≥ 24 hours prior to randomization) will be excluded. During screening (or within 24 hours prior to or after randomization), locally available COVID-19 drugs with antiviral effects (including but not limited to nirmatrelvir/ritonavir, molnupiravir, favipiravir, monoclonal antibodies) will be permitted.
* Other known active viral or bacterial infection at the time of screening, such as influenza and respiratory syncytial virus (RSV). Note: This exclusion does not apply to subjects with stable chronic viral infections, such as chronic hepatitis C virus (HCV) or HIV providing other eligibility criteria are met.
* Receiving dialysis or have known severe renal impairment
* History of severe hepatic impairment (Child-Pugh Class C)
* Known allergy or hypersensitivity to components of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2285 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (202):
- United States (49):
  - Atea Study Site, Kingman, Arizona
  - Atea Study Site, Prescott, Arizona
  - Atea Study Site, Surprise, Arizona
  - Atea Study Site, Tucson, Arizona
  - Atea Study Site, Canoga Park, California
  - Atea Study Site, Fullerton, California
  - Atea Study Site, Inglewood, California
  - Atea Study Site, La Palma, California
  - Atea Study Site, Long Beach, California
  - Atea Study Site, Los Angeles, California
  - Atea Study Site, Sacramento, California
  - Atea Study Site, San Diego, California
  - Atea Study Site, Coral Gables, Florida
  - Atea Study Site, Cutler Bay, Florida
  - Atea Study Site, Doral, Florida
  - Atea Study Site, Hialeah, Florida
  - Atea Study Site, Miami, Florida
  - Atea Study Site, Miami Gardens, Florida
  - Atea Study Site, North Miami Beach, Florida
  - Atea Study Site, Pembroke Pines, Florida
  - Atea Study Site, Pompano Beach, Florida
  - Atea Study Site, Tampa, Florida
  - Atea Study Site, The Villages, Florida
  - Atea Study Site, West Miami, Florida
  - Atea Study Site, West Palm Beach, Florida
  - Atea Study Site, Eatonton, Georgia
  - Atea Study Site, Orland Park, Illinois
  - Atea Study Site, La Vista, Nebraska
  - Atea Study Site, The Bronx, New York
  - Atea Study Site, Chapel Hill, North Carolina
  - Atea Study Site, High Point, North Carolina
  - Atea Study Site, Chickasha, Oklahoma
  - Atea Study Site, Providence, Rhode Island
  - Atea Study Site, Greenville, South Carolina
  - Atea Study Site, Rock Hill, South Carolina
  - Atea Study Site, Carrollton, Texas
  - Atea Study Site, Dallas, Texas
  - Atea Study Site, DeSoto, Texas
  - Atea Study Site, Forney, Texas
  - Atea Study Site, Fort Worth, Texas
  - Atea Study Site, Harlingen, Texas
  - Atea Study Site, Houston, Texas
  - Atea Study Site, Kingwood, Texas
  - Atea Study Site, Lewisville, Texas
  - Atea Study Site, Mesquite, Texas
  - Atea Study Site, San Antonio, Texas
  - Atea Study Site, Splendora, Texas
  - Atea Study Site, Stafford, Texas
  - Atea Study Site, Sugar Land, Texas
- Argentina (12):
  - Atea Study Site, Bahía Blanca, Buenos Aires
  - Atea Study Site, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Atea Study Site, Mar del Plata, Buenos Aires
  - Atea Study Site, Ramos Mejía, Buenos Aires
  - Atea Study Site, San Nicolás de los Arroyos, Buenos Aires
  - Atea Study Site, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Atea Study Site, Córdoba, Córdoba Province
  - Atea Study Site, Rosario, Santa Fe Province
  - Atea Study Site, San Miguel de Tucumán, Tucumán Province
  - Atea Study Site, Ciudad Autonoma de Buenos Aire
  - Atea Study Site, Córdoba
  - Atea Study Site, Santiago del Estero
- Brazil (32):
  - Atea Study Site, Maceió, Alagoas
  - Atea Study Site, Fortaleza, Ceará
  - Atea Study Site, Cachoeiro de Itapemirim, Espírito Santo
  - Atea Study Site, Serra, Espírito Santo
  - Atea Study Site, Vitória, Espírito Santo
  - Atea Study Site, Salvador, Estado de Bahia
  - Atea Study Site, Brasília, Federal District
  - Atea Study Site, Cuiabá, Mato Grosso
  - Atea Study Site, Belo Horizonte, Minas Gerais
  - Atea Study Site, Campina Grande do Sul, Paraná
  - Atea Study Site, Rio de Janeiro, Rio Do Janeiro
  - Atea Study Site, Natal, Rio Grande do Norte
  - Atea Study Site, Passo Fundo, Rio Grande do Sul
  - Atea Study Site, Porto Alegre, Rio Grande do Sul
  - Atea Study Site, Porto Velho, Rondônia
  - Atea Study Site, Blumenau, Santa Catarina
  - Atea Study Site, Florianópolis, Santa Catarina
  - Atea Study Site, Itajaí, Santa Catarina
  - Atea Study Site, Joinville, Santa Catarina
  - Atea Study Site, Barretos, São Paulo
  - Atea Study Site, Bento Gonçalves, São Paulo
  - Atea Study Site, Botucatu, São Paulo
  - Atea Study Site, Campinas, São Paulo
  - Atea Study Site, Ijuí, São Paulo
  - Atea Study Site, Jaú, São Paulo
  - Atea Study Site, Osasco, São Paulo
  - Atea Study Site, Ribeirão Preto, São Paulo
  - Atea Study Site, Santa Catarina, São Paulo
  - Atea Study Site, São José do Rio Preto, São Paulo
  - Atea Study Site, São Paulo, São Paulo
  - Atea Study Site, Valinhos, São Paulo
  - Atea Study Site, Rio de Janeiro
- Canada (2):
  - Atea Study Site, Edmonton, Alberta
  - Atea Study Site, Chicoutimi, Quebec
- Germany (4):
  - Atea Study Site, Munich, Bavaria
  - Atea Study Site, Frankfurt am Main, Hesse
  - Atea Study Site, Berlin
  - Atea Study Site, Hamburg
- India (16):
  - Atea Study Site, Hyderabad, Andhra Pradesh
  - Atea Study Site, Nellore, Andhra Pradesh
  - Atea Study Site, Visakhapatnam, Andhra Pradesh
  - Atea Study Site, Nellore, Andhra Prasesh
  - Atea Study Site, Ahmedabad, Gujarat
  - Atea Study Site, Gotri, Gujarat
  - Atea Study Site, Surat, Gujarat
  - Atea Study Site, Faridabad, Haryana
  - Atea Study Site, Bangalore, Karnataka
  - Atea Study Site, Bengaluru, Karnataka
  - Atea Study Site, Dombivali, Maharashtra
  - Atea Study Site, Nashik, Maharashtra
  - Atea Study Site, Pune, Maharashtra
  - Atea Study Site, New Delhi, National Capital Territory of Delhi
  - Atea Study Site, Jaipur, Rajasthan
  - Atea Study Site, Chennai, Tamil Nadu
- Japan (16):
  - Atea Study Site, Fukuoka, Fukuoka
  - Atea Study Site, Kasuga, Fukuoka
  - Atea Study Site, Kitakyushu, Fukuoka
  - Atea Study Site, Fukuoka, Fukuoka City
  - Atea Study Site, Sapporo, Hokkaido
  - Atea Study Site, Himeji, Hyōgo
  - Atea Study Site, Tsuchiura, Ibaraki
  - Atea Study Site, Kanazawa, Ishikawa-ken
  - Atea Study Site, Fujisawa, Kanagawa
  - Atea Study Site, Kamakura, Kanagawa
  - Atea Study Site, Izumisano, Osaka
  - Atea Study Site, Toda, Saitama
  - Atea Study Site, Uozu, Toyama
  - Atea Study Site, Chiba
  - Atea Study Site, Fukuoka
  - Atea Study Site, Okayama
- Latvia (2):
  - Atea Study Site, Daugavpils
  - Atea Study Site, Riga
- Mexico (13):
  - Atea Study Site, Saltillo, Coahuila
  - Atea Study Site, Torreón, Coahuila
  - Atea Study Site, Guadalajara, Jalisco
  - Atea Study Site, Mexico City, Mexico City
  - Atea Study Site, Monterrey, Nuevo León
  - Atea Study Site, Querétaro City, Querétaro
  - Atea Study Site, Cancún, Quintana Roo
  - Atea Study site, San Luis Potosí City, San Luis Potos
  - Atea Study Site, Yucatán, Yucatán
  - Atea Study Site, Chihuahua City
  - Atea Study Site, Oaxaca City
  - Atea Study Site, Puebla City
  - Atea Study Site, Veracruz
- Netherlands (3):
  - Atea Study Site, The Hague
  - Atea Study Site, Utrecht
  - Atea Study Site, Zwijndrecht
- Pakistan (4):
  - Atea Study Site, Islamabad
  - Atea Study Site, Karachi
  - Atea Study Site, Lahore
  - Atea Study Site, Rawalpindi
- Philippines (6):
  - Atea Study Site, Baguio City, Cordillera
  - Atea Study Site, Tacloban City, Leyte
  - Atea Study Site, Ermita, Manila
  - Atea Study Site, San Fernando City, Pampanga
  - Atea Study Site, Iloilo City
  - Atea Study Site, Mandaluyong
- Romania (8):
  - Atea Study Site, Baloteşti
  - Atea Study Site, Bucharest
  - Atea Study Site, Constanța
  - Atea Study Site, Craiova
  - Atea Study Site, Oradea
  - Atea Study Site, Sibiu
  - Atea Study Site, Suceava
  - Atea Study Site, Timișoara
- South Africa (8):
  - Atea Study Site, East London, Eastern Cape
  - Atea Study Site, Johannesburg, Gauteng
  - Atea Study Site, Pretoria, Gauteng
  - Atea Study Site, Randburg, Gauteng
  - Atea Study Site, Thabazimbi, Limpopo
  - Atea Study Site, Kimberley, Northern Cape
  - Atea Study Site, Cape Town, Western Cape
  - Atea Study Site, Plettenberg Bay, Western Cape
- Spain (6):
  - Atea Study Site, Badalona, Barcelona
  - Atea Study Site, Centelles, Barcelona
  - Atea Study Site, Marbella, Malaga
  - Atea Study Site, Málaga, Malaga
  - Atea Study Site, Barcelona
  - Atea Study Site, Madrid
- Sweden (2):
  - Atea Study Site, Solna
  - Atea Study Site, Umeå
- Tunisia (6):
  - Atea Study Site, La Marsa
  - Atea Study Site, Monastir
  - Atea Study Site, Montfleury
  - Atea Study Site, Sfax
  - Atea Study Site, Sousse
  - Atea Study Site, Tunis
- Turkey (Türkiye) (9):
  - Atea Study Site, Ankara
  - Atea Study Site, Antalya
  - Atea Study Site, Bursa
  - Atea Study SIte, Denizli
  - Atea Study Site, Istanbul
  - Atea Study Site, Izmir
  - Atea Study SIte, Kayseri
  - Atea Study Site, Samsun
  - Atea Study Site, Yenimahalle
- United Kingdom (4):
  - Atea Study Site, Exeter, Devon
  - Atea Study Site, Plymouth, Devon
  - Atea Study Site, London, Greater London
  - Atea Study Site, Castleford, West Yourkshire

RESULTS

PARTICIPANT FLOW:
Groups:
- BEM - SCO Stratum; PBO - SCO Stratum: Supportive Care Only (SCO) Stratum are subjects who did not receive any treatment with direct SARS-CoV-2 antiviral activity in parallel with study drug (BEM or placebo (PBO)).
- BEM - Combo Stratum; PBO - Combo Stratum: Combination (Combo) Stratum are subjects who did receive treatment with direct SARS-CoV-2 antiviral activity in parallel with study drug (BEM or placebo (PBO)).
Period: Through Day 29
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Started | 1104 | 1107 | 38 | 36
Completed | 1073 | 1087 | 37 | 35
Not Completed | 31 | 20 | 1 | 1
Period: Day 30 Through Day 60
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Started | 1073 | 1087 | 37 | 35
Completed | 1071 | 1083 | 37 | 35
Not Completed | 2 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included subjects who received >= 1 dose of study drug and had >= 1 positive SARS-CoV-2 result through Day 5.
Groups:
- Total: Total of all reporting groups
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum | Total
Number analyzed (Participants) | 1022 | 1033 | 36 | 34 | 2125
Age, Customized [Count of Participants; unit: Participants]
  18-49 years | 28 | 30 | 1 | 2 | 61
  50-64 years | 429 | 432 | 13 | 13 | 887
  65-79 years | 486 | 487 | 18 | 17 | 1008
  >= 80 years | 79 | 84 | 4 | 2 | 169
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 613 | 634 | 18 | 22 | 1287
  Male | 409 | 399 | 18 | 12 | 838
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 861 | 875 | 16 | 18 | 1770
  Not Hispanic or Latino | 123 | 131 | 19 | 16 | 289
  Unknown or Not Reported | 38 | 27 | 1 | 0 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 11 | 1 | 0 | 20
  Asian | 68 | 55 | 3 | 1 | 127
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 73 | 73 | 3 | 2 | 151
  White | 867 | 882 | 24 | 28 | 1801
  More than one race | 1 | 4 | 0 | 0 | 5
  Unknown or Not Reported | 5 | 8 | 5 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Hospitalized for Any Cause or Died Due to Any Cause
Time Frame: Day 1 through Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Number analyzed (Participants) | 1022 | 1033 | 36 | 34
Participants | 7 | 2 | 0 | 0
Statistical Analysis 1: Comparison: BEM - SCO Stratum vs PBO - SCO Stratum; Test type: Superiority; p = 0.954, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Subjects Hospitalized Due to COVID-19 or Died Due to Any Cause
Time Frame: Day 1 through Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Number analyzed (Participants) | 1022 | 1033 | 36 | 34
Participants | 4 | 2 | 0 | 0

3. Secondary Outcome: Percentage of Subjects Who Died Due to Any Cause
Time Frame: Day 1 through Day 29; Day 1 through Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Number analyzed (Participants) | 1022 | 1033 | 36 | 34
Participants
  Through Day 29 | 2 | 1 | 0 | 0
  Through Day 60 | 3 | 1 | 0 | 0

4. Secondary Outcome: Percentage of Subjects With COVID-19-related Complications
Time Frame: Day 1 through Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Number analyzed (Participants) | 1022 | 1033 | 36 | 34
Participants | 3 | 4 | 0 | 0

5. Secondary Outcome: Percentage of Subjects With COVID-19-medically Attended Visits (Hospitalization, Emergency Room (ER) Visit, Urgent Care Visit, Physician's Office Visit, or Telemedicine Visit) or Who Died Due to Any Cause
Time Frame: Day 1 through Day 29; Day 1 through Day 60
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Number analyzed (Participants) | 1022 | 1033 | 36 | 34
Participants
  Through Day 29 | 7 | 11 | 1 | 0
  Through Day 60 | 8 | 12 | 1 | 0

6. Secondary Outcome: Percentage of Subjects With COVID-19 Symptom Relapse
Time Frame: Day 1 through Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Number analyzed (Participants) | 1022 | 1033 | 36 | 34
Participants | 272 | 265 | 13 | 12

7. Secondary Outcome: Percentage of Subjects With Viral Load Rebound
Time Frame: Day 1 through Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
Number analyzed (Participants) | 1022 | 1033 | 36 | 34
Participants | 79 | 102 | 4 | 5

ADVERSE EVENTS:
Time Frame: Through Day 60
Description: Serious adverse events were collected through Day 60. Non-serious adverse events were collected through Day 29.
  Systematic Assessment: Regular investigator assessment at each study visit.
Groups:
- BEM - SCO Stratum; PBO - SCO Stratum: Supportive Care Only (SCO) Stratum are subjects who did not receive any treatment with direct SARS-CoV-2 antiviral activity in parallel with study drug (BEM or placebo (PBO)).
  Safety population includes all subjects who received at least one dose of the study drug (BEM or PBO).
- BEM - Combo Stratum; PBO - Combo Stratum: Combination (Combo) Stratum are subjects who did receive treatment with direct SARS-CoV-2 antiviral activity in parallel with study drug (BEM or placebo (PBO)).
  Safety population includes all subjects who received at least one dose of the study drug (BEM or PBO).
Arm/Group | BEM - SCO Stratum | PBO - SCO Stratum | BEM - Combo Stratum | PBO - Combo Stratum
All-Cause Mortality (participants affected / at risk) | 3/1093 | 1/1103 | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 9/1093 | 2/1103 | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 39/1093 | 35/1103 | 6/37 | 9/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEM - SCO Stratum (N=1093) | PBO - SCO Stratum (N=1103) | BEM - Combo Stratum (N=37) | PBO - Combo Stratum (N=36)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BEM - SCO Stratum (N=1093) | PBO - SCO Stratum (N=1103) | BEM - Combo Stratum (N=37) | PBO - Combo Stratum (N=36)
Diarrhoea (Gastrointestinal disorders) | 24 | 24 | 4 | 3
Nausea (Gastrointestinal disorders) | 11 | 10 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 4 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 2
Dysguesia (Nervous system disorders) | 0 | 0 | 3 | 1

LIMITATIONS AND CAVEATS:
The study was originally designed based on available epidemiological data at the time including an assumed hospitalization or death rate in the range of 3% to 6%. The overall global decline in hospitalizations during the study ultimately blunted the ability to detect the efficacy of BEM.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication or presentation of data from individual study centers is subject to prior review by the Sponsor. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT05629962/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT05629962/SAP_001.pdf